CLINICAL TRIAL: NCT05494645
Title: Exparel Use in Peripheral Nerve Blocks and Local Infiltration for Foot and Ankle Surgery: A Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: SLRI-2022-24
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-07

CONDITIONS: Pain, Postoperative; Pain, Acute Postoperative; Ankle Fractures; Ankle Injuries and Disorders
Keywords: liposomal bupivacaine; ankle surgery; postoperative pain; regional nerve block
MeSH Terms: conditions — Pain, Postoperative; Ankle Fractures; Ankle Injuries; Disease | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: patient is blinded to study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Peripheral Nerve Block Without Exparel (Active Comparator): Lower extremity peripheral nerve block without Exparel: 0.25-0.5% bupivacaine
  Interventions: Drug: Peripheral Nerve Block
- Peripheral Nerve Block with Exparel (Experimental): Liposomal bupivicaine administered for peripheral nerve block: mixed with 0.25-0.5% bupivacaine
  Interventions: Drug: Exparel
- Local Infiltration of Exparel (Experimental): Liposomal bupivicaine administered by surgeon intra-operatively in field block, mix with 0.25% bupivacaine
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Exparel — Liposomal bupivicaine
  Other Names: Liposomal bupivicaine
  Arms: Local Infiltration of Exparel; Peripheral Nerve Block with Exparel
Drug: Peripheral Nerve Block — Peripheral nerve block without Exparel
  Other Names: marcaine, bupivicaine
  Arms: Peripheral Nerve Block Without Exparel

SUMMARY:
Liposomal Bupivacaine (Exparel) has been recently studied as the active agent utilized in various nerve block. Due to its liposomal form allowing for extended delivery, Exparel has been used in various peri-operative nerve blocks among multiple orthopaedic specialties in hopes of achieving improved pain control and decreased opioid use. This study compares the efficacy and effect on opioid use of peripheral nerve blocks and local infiltration with and without Exparel in patients undergoing foot and ankle surgery.

DETAILED DESCRIPTION:
three study groups: A - surgeon infiltrates with exparel on site of surgery; B - anesthesia provides a regional nerve block (popliteal/adductor blocks) with plain local anesthetic (bupivacaine); C - anesthesia provides a regional nerve block (popliteal/adductor) with Exparel/bupivacaine mix. Follow up occurs on postop day 4 via phone call to patient. Measured outcomes include opioid consumption in post anesthesia care unit phase (oral morphine equivalents), block duration, number of opioid pills used by postop day 4, oral morphine equivalent consumption by postop day 4.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective orthopaedic foot and ankle surgery at a single institution
* English speaking
* Able to provide consent to surgery and study participation

Exclusion Criteria:

* Non-elective or emergent foot and ankle surgery
* Non-english speaking
* Does not possess medical decision making capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of block | 3 Months

SECONDARY OUTCOMES:
number of opioid pills used by postoperative day # 4 | 3 months
PROMIS Scores | 3 months
oral morphine equivalent use by postoperative day 4 | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna Ng-Pellegrino, Principal Investigator — St. Luke's Hospital and Health Network, Pennsylvania
Locations (1):
- St. Luke's University Health Network, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No